CLINICAL TRIAL: NCT04717687
Title: Étude Pilote de l'évaluation de la Technique de l'électroporation irréversible Dans le Cholangiocarcinome Infiltrant périhilaire
Brief Title: Pilot Study on the Evaluation of Irreversible Electroporation Technique in Infiltrating Perihilar Cholangiocarcinoma
Acronym: HOPE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: Poitiers University Hospital (Other)
Collaborators: Sport & Collection 2019 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOPE
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Cholangiocarcinoma; Interventional Imaging
Keywords: Cholangiocarcinoma; Irreversible electroporation; Interventional radiology
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrodes (Experimental): Electrodes
  Interventions: Procedure: Irreversible electroporation

INTERVENTIONS:
Procedure: Irreversible electroporation — Device: NanoKnife The aim of the treatment is to surround the tumour with two to six needles and to deliver a very high voltage current (3000 volts in 70 to 80 microseconds pulses) by a generator synchronized with an electrocardiogram.

SUMMARY:
The aim of the study is to evaluate the feasibility of irreversible electroporation in the treatment of locally advanced cholangiocarcinoma. This technique would allow to treat the unresectable part of the tumor to make it more accessible for a secondary surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Patient with infiltrating cholangiocarcinoma of the gallstone convergence considered as unresectable on the pre-operative imaging data performed during the month preceding inclusion, and in multidisciplinary consultation meeting specialised in digestive oncology
* Histologically (or cytologically) proven tumor of less than 4 cm of the largest diameter
* World Health Organization Performance Index 0 or 1
* No history of other cancer, except baso-cellular skin carcinoma or epidermoid cervix cancer or any other cancer in complete remission for more than 3 years
* No prior radiotherapy for cholangiocarcinoma
* Biological analyses performed during the month preceding inclusion : hepatic enzymes (AST and ALT <3N), preserved renal function (creatinine clearance according to Modification of the Diet in Renal Disease >50ml/min); bilirubin <3N; bile drainage must be correct with a bilirubin below 3N , with or without drainage/prothesis, hemoglobin >9g/dL, leucocytes >3500/mm3, platelets >75000/mm3, prothrombin rate >70%
* Signature of the informed consent

Exclusion Criteria:

* Cholangiocarcinoma of more than 4cm diameter or resectable according tio the imaging data
* Severe and/or uncontrolled (cardiac, pulmonary, renal, liver decompensation...) visceral failure, in the 6 months preceding the study
* Visceral metastases or peritoneal carcinosis
* History of cancers except if remission for more than 3 years, in-situ cancer, epidermoid or baso-cellular cancer
* Metal biliary prothesis non extractable
* Patient with history of epileptic events
* History of myocard infarction for less than 6 months
* Unstabilised coronary disease for at least 6 months
* Cardiac rhythm trouble or QT space above 550ms without treatment
* Patient eligible to liver transplant
* Patient naive of chemiotherapy
* Patient with a pacemaker, an implanted automatic defibrillator or an automatic electronic device or an electronic device with metal pieces
* Patient with contra-indication to the use of NanoKnife system
* History of hypersensitivity to gadolinium or to iodized contrast product not allowing a suitable radiologic monitoring
* Refusal or language or psychic incapacity to sign the informed consent
* Subject who cannot submit to the constraints of the protocol (subjects for which an MRI or a scan is contra-indicated, claustrophobic subjects, non cooperative or not able to come to the follow-up visits)
* Concomitant participation to another study
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, adults under legal protection.
* Women at age to procreate and not using effective contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The success rate of the technique, being the realisation of the irreversible electroporation. | At Day 0
  The study will be considered positive if the success rate is above 90% and the complication rate below or equal to 30%